CLINICAL TRIAL: NCT00197106
Title: A Multicentre, Randomised, Double-blind, Parallel Group Study to Compare the Efficacy and Safety of Salmeterol/Fluticasone Propionate Combination Product (Seretide®) 50/100 mcg With Fluticasone Propionate (Flixotide® ) 200 mcg, Both Delivered Twice Daily Via the DISKUS Inhaler, in the Treatment of Children Aged 6-12 Years With Symptomatic Asthma
Brief Title: Treatment Of Symptomatic Asthma In Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAM101667
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Results first posted 2009-12-14 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2012-04

CONDITIONS: Asthma
Keywords: salmeterol/fluticasone combination; Asthma; bronchial hyperresponsiveness; Children; symptom control
MeSH Terms: conditions — Asthma; Bronchial Hyperreactivity | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Salmeterol/ fluticasone propionate Diskus® inhaler 50/100 mcg (Active Comparator): Salmeterol/ fluticasone propionate Diskus® inhaler 50/100 mcg
  Interventions: Drug: Salmeterol/ fluticasone propionate Diskus® inhaler 50/100 mcg
- fluticasone propionate 2 x 100 mcg (Other): fluticasone propionate 2 x 100 mcg
  Interventions: Drug: fluticasone propionate 2 x 100 mcg

INTERVENTIONS:
Drug: Salmeterol/ fluticasone propionate Diskus® inhaler 50/100 mcg — comparator
  Arms: Salmeterol/ fluticasone propionate Diskus® inhaler 50/100 mcg
Drug: fluticasone propionate 2 x 100 mcg — comparator
  Other Names: Salmeterol/ fluticasone propionate Diskus® inhaler 50/100 mcg
  Arms: fluticasone propionate 2 x 100 mcg

SUMMARY:
This study is being conducted to investigate whether in childhood salmeterol/ fluticasone propionate 50/100 bd delivered via the Diskus® inhaler and fluticasone propionate 200 mcg bd delivered via the Diskus® inhaler are non- inferior in terms of symptom control. Additionally we aim to show that salmeterol/ fluticasone propionate 50/100 bd is at least as good in terms of lung function improvement and bronchial hyperreactivity and enables a steroid-sparing management of asthma in children.

DETAILED DESCRIPTION:
A multicentre, randomised, double blind, parallel group study to compare the efficacy and safety of Salmeterol/Fluticasone propionate combination product (Seretide®) 50/100mcg with Fluticasone propionate (Flixotide®) 200mcg, both delivered twice daily via the DISKUS inhaler, in the treatment of children aged 6-12 years with symptomatic asthma.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects aged 6-12 years (inclusive)
* A female is eligible to enter and participate in the study if she is:

of non-child-bearing potential; OR of child-bearing potential, but not lactating and pregnant. She declares that it is not probable that she will become pregnant during the study (a pregnancy test can be performed at the investigators discretion)

* Subjects with a documented history of asthma for at least 6 months
* Subjects with a documented history of BHR within 12 months prior to inclusion or BHR on visit 1 (PD20 methacholine < 150 mcg or an equivalence for histamine)
* Subjects who have received BDP, budesonide up to 100-200 mcg bd or fluticasone propionate at a dose of up to 125 mcg bd for at least 4 weeks before the start of the run-in period.
* Subjects who are able to use a electronic peakflow /FEV1 meter (PIKO-1)
* Subjects who have a normal length SD score between -2SD and +2SD
* Subjects who are able to use a Diskus inhaler
* Subjects who are able to perform reproducible lung function tests at visit 1 (variation FEV1 < 5% between the two best measurements)
* Subjects and their guardians, who have given written informed consent to participate in the study
* Subjects or their parent/ guardian who are able to understand and complete a DRC. The DRC may be completed by a parent/guardian if the subject is unable to do this him/ herself
* Subjects able to use Ventolin on an 'as required for symptoms' basis

Exclusion criteria:

* Subjects who have been hospitalised for their asthma within 4 weeks of visit 1
* Subjects who had an acute upper respiratory tract infection within 2 weeks or a lower respiratory tract infection within 4 weeks prior to visit 1
* Subjects who received oral, parental or depot corticosteroids within 4 weeks prior to visit 1
* Subjects who have a known respiratory disorder other than asthma and/or systemic/thoracic abnormalities which influence normal lung function
* Subjects with a disorder that affects growth (e.g. Turner's syndrome)
* Subjects who have received any investigational drugs within 4 weeks of visit 1
* Subjects with a known or suspected hypersensitivity to inhaled steroids, β2-agonists or lactose
* Subjects who use any medication that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4, including ritonavir and ketoconazole
* Subjects who concurrently participate in another clinical study
* Subjects who have previously been randomised in this trial

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2005-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- Netherlands (18):
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Gouda
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Helmond
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Sittard
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Veldhoven
  - GSK Investigational Site, Zwolle

REFERENCES:
- [Derived] Vaessen-Verberne AA, van den Berg NJ, van Nierop JC, Brackel HJ, Gerrits GP, Hop WC, Duiverman EJ; COMBO Study Group. Combination therapy salmeterol/fluticasone versus doubling dose of fluticasone in children with asthma. Am J Respir Crit Care Med. 2010 Nov 15;182(10):1221-7. doi: 10.1164/rccm.201002-0193OC. Epub 2010 Jul 9. PMID 20622031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were eligible to enter the run-in period if they had a documented clinical history of asthma with hyperresponsiveness. Only participants who were symptomatic after this period were eligible to be enrolled into the study and were randomized into either the Salmeterol/Fluticasone propionate (FP) 50/100 mcg plus placebo or FP groups.
Pre-assignment Details: 257 participants started the run-in phase of the study, and 99 of these did not meet the inclusion criteria to be entered into the treatment phase. Only baseline characteristics for the 158 participants meeting the inclusion criteria and randomized to either salmeterol/fluticasone propionate 50/100 mcg BID or fluticasone 200 mcg BID are provided.
Groups:
- Fluticasone Propionate (FP) 100 mcg: Fluticasone propionate (FP) 100 mcg (micrograms) twice daily (BID) via DISKUS inhaler
- Salmeterol/FP 50/100 mcg Plus Placebo: One puff Salmeterol/FP 50/100 mcg plus one puff placebo (matching one puff of FP in the 200 mcg group) BID via DISKUS inhaler
- FP 200 mcg: FP 200 mcg (delivered as two 100 mcg puffs) BID via DISKUS inhaler
Period: 4-Week Run-In Period
Arm/Group | Fluticasone Propionate (FP) 100 mcg | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Started | 257 | 0 | 0
Completed | 158 | 0 | 0
Not Completed | 99 | 0 | 0
Not completed — Did not meet entry criteria | 99 | 0 | 0
Period: Overall Treatment Period
Arm/Group | Fluticasone Propionate (FP) 100 mcg | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Started | 0 | 78 | 80
Completed | 0 | 77 | 74
Not Completed | 0 | 1 | 6
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Salmeterol/FP 50/100 mcg Plus Placebo: Salmeterol/FP 50/100 mcg plus placebo BID via DISKUS inhaler
- FP 200 mcg: FP 200 mcg BID via DISKUS inhaler
- Total: Total of all reporting groups
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg | Total
Number analyzed (Participants) | 78 | 80 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (1.8) | 9.3 (1.9) | 9.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 31 | 67
  Male | 42 | 49 | 91
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 73 | 75 | 148
  Mixed | 4 | 3 | 7
  African-American | 0 | 1 | 1
  African | 1 | 1 | 2
Asthma duration [Mean (Standard Deviation); unit: years] — Mean asthma duration before enrollment in study
  years | 5.7 (3.1) | 5.5 (3.0) | 5.6 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Symptom-free Days During the Last 10 Weeks of the Treatment Period
Description: Asthma symptom-free days are defined as days (24 hour period) with no symptoms, as recorded in the participant's diary.
Time Frame: Last 10 weeks of the treatment period (Weeks 16-26)
Population: Per protocol (PP) population: participants of the Intent-to-Treat (ITT) Population (participants who had taken at least one dose of study medication) who completed the study without any major protocol violations
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 73 | 76
percentage of days | 50.45 (33.52) | 49.75 (35.77)
Statistical Analysis 1: Comparison: Salmeterol/FP 50/100 mcg Plus Placebo vs FP 200 mcg; Test type: Non-Inferiority or Equivalence — Non-inferiority is considered to be shown if the upper limit of the one-sided 95% confidence interval of the difference uflixotide-useretide does not exceed +15% (uflixotide-useretide represent the mean percentages of asthma symptom-free days of the two respective treatment groups); p = 0.63, Repeated Measurements Anal. of Variance; Anal. = Analysis; Adjusted difference = 2.6, 95% CI [-8.1 to 13.4]

2. Secondary Outcome: Percentage of Symptom-free Days During the Entire Treatment Period
Description: Asthma symptom-free days are defined as days (24 hour period) with no symptoms, as recorded in the participant's diary
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 73 | 76
percentage of days
  Baseline | 22.78 (25.30) | 23.06 (25.23)
  0-6 weeks | 31.58 (31.34) | 31.50 (29.73)
  6-16 weeks | 44.60 (34.67) | 45.24 (34.58)
  16-26 weeks | 50.45 (33.52) | 49.75 (35.77)

3. Secondary Outcome: Mean Change From Baseline in Percentage Predicted Forced Expiratory Volume in One Second (FEV1) at Week 26
Description: Change from Baseline was calculated as the Week 26 value minus the Baseline value. The percentage predicted FEV1 is defined as the volume of air that can be forced out in one second after taking a deep breath and is corrected for the FEV1 value corresponding with the same age.
Time Frame: Baseline and Week 26
Population: Per protocol (PP) population: participants of the Intent-to-Treat (ITT) Population (participants who had taken at least one dose of study medication) who completed the study without any major protocol violations. At baseline there were 6 missing data and 4 improper testings that could not be used in the analysis.
Measure: Mean (Standard Deviation); unit: percent predicted change
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 61 | 61
percent predicted change | 102.5 (14.2) | 103.0 (15.3)

4. Secondary Outcome: Mean Change From Baseline in Forced Vital Capacity (FVC) at Week 26
Description: Change from Baseline was calculated as the Week 26 value minus the Baseline value. Forced vital capacity is defined as the maximum volume of air that can be forcibly expired from the lungs and is calculated by use of spirometry. The spirometry test is performed by using a device called a spirometer, which measures the amount of air one can blow out maximally. Generally, the participant is asked to take the deepest breath they can, and then exhale into the sensor as hard as possible, for as long as possible. The test is normally repeated three times to ensure reproducibility.
Time Frame: Baseline and Week 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 61 | 61
liters | 2.28 (0.62) | 2.28 (0.59)

5. Secondary Outcome: Mean Change From Baseline in Midexpiratory Flow (MEF 50) at Week 26
Description: Change from Baseline was calculated as the Week 26 value minus the Baseline value. MEF 50 is defined as maximum expiratory flow rate at 50% of vital capacity. Vital capacity is the maximum amount of air that a person can expel from the lungs after first filling the lungs to their maximum extent. Midexpiratory flow was calculated by use of spirometry. The test is normally repeated at least three times in order to ensure reproducibility.
Time Frame: Baseline and Week 26
Population: Per protocol (PP) population: participants of the Intent-to-Treat (ITT) Population (participants who had taken at least one dose of study medication) who completed the study without any major protocol violations. For some participants, the data for the MEF 50 measurements are missing, resulting in a smaller number of participants analyzed.
Measure: Mean (Standard Deviation); unit: liters/second
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 57 | 57
liters/second | 2.28 (0.67) | 2.19 (0.72)

6. Secondary Outcome: Geometric Means of Nitric Oxide (NO) at Week 26
Description: Geometric mean values of NO at week 26 were compared using ANCOVA with adjustment for baseline value of NO, age, gender and center. Analysis of covariance (ANCOVA) is a general linear model with one continuous outcome variable (quantitative) and one or more factor variables.
Time Frame: Baseline and Week 26
Population: Per protocol (PP) population: participants of the Intent-to-Treat (ITT) Population (participants who had taken at least one dose of study medication) who completed the study without any major protocol violations and completed two NO measurements (Baseline and Week 26)
Measure: Geometric Mean (Full Range); unit: parts per billion
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 27 | 31
parts per billion | 8.6 [1.9 to 64.0] | 10.0 [1.8 to 51.6]

7. Secondary Outcome: Percent Change From Baseline in RINT Measurements at Week 26
Description: Change from Baseline was calculated as the Week 26 value minus the Baseline value. Interrupter respiratory resistance (RINT) measurements were calculated by a combined analysis for relation between change from baseline and occurrence of the endpoint. RINT is a technique that is used for evaluating lung function in poorly collaborating patients (e.g., small children). The measurement is performed during tidal breathing (normal breathing) instead of during maximal expiration, as is done by a spirometry test.
Time Frame: Baseline and Week 26
Population: PP Population: Intent-to-Treat (ITT) Population participants who completed the study without any major protocol violations and completed two NO measurements (Baseline and Week 26). For some participants, the data for the RINT measurement are missing, either at Baseline or at Week 26. As a result, fewer subjects have been included in the analysis.
Measure: Number; unit: percent
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 57 | 57
percent | -9.1 | -9.9

8. Secondary Outcome: Number of Asthma Exacerbations Per Treatment Group at Week 26
Description: An exacerbation is defined as a worsening of the asthma complaints (commonly referred to as an asthma attack) and is reported by the participant experiencing the event. An exacerbation was verified by the use of asthma rescue medication.
Time Frame: Week 26
Population: Intent-to-Treat (ITT) Population (participants who had taken at least one dose of study medication)
Measure: Number; unit: number of exacerbations
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 80 | 78
number of exacerbations | 10 | 7

9. Secondary Outcome: Mean Change From Baseline in Provocation Dose (PD20) Causing a 20% Fall in FEV1 at Week 26
Description: PD20 was calculated by using increasing dosages of methacholine. The dosage that caused a 20% fall in FEV1 was used for analysis. The presented data are ratios (month 6/Baseline) of geometric mean PD20 values.
Time Frame: Baseline and Week 26
Population: Per protocol (PP) population: participants of the Intent-to-Treat (ITT) Population (participants who had taken at least one dose of study medication) who completed the study without any major protocol violations. From this population, only participants who had measurements at both baseline and Week 26 have been used for analysis.
Measure: Log Mean (95% Confidence Interval); unit: ratio
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 65 | 61
ratio | 2.7 [1.05 to 6.7] | 1.5 [0.7 to 2.9]

10. Secondary Outcome: Bronchial Hyperresponsiveness With PD20 AMP in Selected Centres
Description: Bronchial hyperresponsiveness with PD20 AMP in selected centres was not analyzed, as this outcome measure was removed in a protocol amendment.
Time Frame: 26 weeks
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Daily FEV1 and PEF Via the Electronic Peak Flow/FEV1 Meter (PIKO-1)
Description: Daily FEV1 and PEF via the electronic pea kflow/FEV1 meter (PIKO-1) was not assessed because data from the peak flow meters could not be used for analysis.
Time Frame: 26 weeks
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Frequency of Asthma Exacerbations (Discriminated on Severity)
Description: The frequency of asthma exacerbations (discriminated on severity) was not analyzed because of the low overall frequency.
Time Frame: 26 weeks
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Cumulative Number of Symptom-free Weeks Until the End of Treatment
Description: This outcome measure was not analyzed due to different insights after protocol finalization; it has become clear that the definition of good and maximal controlled weeks is not very distinctive and can therefore actually not be used.
Time Frame: 26 weeks
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Weekly Percentage of Participants With 'Good Controlled Weeks' and 'Maximal Controlled Weeks'
Description: as for outcome 13
Time Frame: 26 weeks
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Time to Asthma Control, Defined as the Time to First 'Good Controlled Week' or 'Maximum Controlled Week'
Description: as for outcome 13
Time Frame: 26 weeks
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Salmeterol/FP 50/100 mcg Plus Placebo | FP 200 mcg
Serious Adverse Events (participants affected / at risk) | 2/78 | 3/80
Other Adverse Events (participants affected / at risk) | 40/78 | 44/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Salmeterol/FP 50/100 mcg Plus Placebo (N=78) | FP 200 mcg (N=80)
Worsening of asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Reactive arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Salmeterol/FP 50/100 mcg Plus Placebo (N=78) | FP 200 mcg (N=80)
Common cold (Respiratory, thoracic and mediastinal disorders) | 28 | 17
Headache (Nervous system disorders) | 14 | 21
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.